CLINICAL TRIAL: NCT00179907
Title: A Phase I/II Study of Reirradiation for Recurrent Pediatric Brain and Spinal Cord Tumors and Primary Glioblastoma Multiforme Using the Photon Radiosurgery System
Brief Title: A Phase I/II Study of the Photon Radiosurgery System
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: Photoelectron Corporation (Unknown)
Responsible Party: Principal Investigator, Stewart Goldman, Attending, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNS 0201
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2015-03-02 (Estimated); Status verified 2015-02

CONDITIONS: Brain Tumor, Recurrent; Glioblastoma Multiforme
MeSH Terms: conditions — Brain Neoplasms; Glioblastoma

INTERVENTIONS:
Procedure: Photon Radiosurgery System (Intrabeam) — In this study we had intended to perform a similar dose escalation study with doses ranging from 10-19 Gy, 10-16 Gy and 10 - 14 Gy for tumors < 20 mm, 21-25 mm and 26-40 mm respectively

SUMMARY:
The standard treatment for children with brain tumors is surgical removal of the tumor followed by radiation to the brain and chemotherapy (medicines) given to shrink any remaining tumor or to prevent tumor from growing back. There are very few treatment options available for children whose brain tumor grows back after receiving radiation treatment. There is a greater risk of complications and side effects when the brain is repeatedly treated with external radiation. The side effects of repeat radiation treatment are dependent on the amount of the brain that is radiated. Radiation given with PRS during surgery is focused to the specific area of the brain where the tumor is located. Therefore, the area of the brain affected by the radiation is smaller. It is hoped that this targeted radiation will lessen the side effects to the normal brain that is not affected by the tumor. It is also hoped that a lower occurrence of side effects will increase the quality of life of children with brain tumors.

The optimal dose of targeted radiation is not known. Therefore, increasing doses will be given to treat different patients, starting with the lowest possible dose. The amount of radiation to be given will depend on whether or not your child received prior radiation therapy and where the tumor is located. The groups of patients will first be divided into 2 groups: Group A, who are those who received radiation as part of their prior treatment, and Group B, who are those who did not receive any radiation treatment. Each group will be then divided again into 2 groups depending on the location of the tumor. In each group, if the lowest dose is well-tolerated with only minimal side effects by 3 patients, then the next higher dose will be given to the next 3 patients.

The purposes of this research are:

* To evaluate the potential side effects of a single high dose of x-rays using the Photon Radiosurgery System (PRS) given to a small area of the brain.
* To determine the maximum dose of targeted radiation that can be safely given to brain tumors with the fewest side effects.
* To see how well this treatment works for children with recurrent brain tumors and newly-diagnosed glioblastoma multiforme.

DETAILED DESCRIPTION:
Central nervous system tumors account for approximately 20% of all childhood neoplasms. The treatment modalities used in the primary management of brain tumors are surgery, radiation therapy and chemotherapy. In recent years, considerable progress has been made in each of these therapeutic approaches. In spite of these advancements local tumor recurrence continues to be an important reason for treatment failure in these children. The local tumor recurrence rate varies according to the primary tumor type, treatment technique and tumor-stage at initial presentation. After conventional treatment, the local tumor recurrence rate ranges from 10% - 40% in tumors like medulloblastoma, craniopharyngioma, ependymoma and low-grade gliomas . However in aggressive tumors like glioblastoma multiforme the tumor recurrence rate in spite of the best modern treatments remains at 80-100%.

Radiation therapy has always played a key role in the management of adult and pediatric brain tumors. There has been considerable interest in treating brain tumors using stereotactic radiosurgery (SRS) using the Gamma knife or Linear accelerator and stereotactic radiotherapy (SRT). The goal of stereotactic treatment is to deliver a high dose of radiation with high geometric precision to a discrete tumor located in the brain. This is accomplished by the use of rigid immobilization skull frames and CT / MRI information for treatment planning and tumor targeting. Presently there are several therapeutic options available for children with recurrent brain tumors. Reirradiation has been employed in recurrent gliomas, medulloblastomas and ependymomas with stereotactic radiosurgery stereotactic radiation and brachytherapy . Following reirradiation, tumor control rates of 50-70% have been obtained. The radiosurgery doses used in children with radiation recurrent tumors have ranged from 10-24 Gy. The reirradiation has been generally well tolerated with retreatment complications like transient edema, cranial neuropathy or radiation necrosis observed in 10-15% of children. The results with high dose chemotherapy and bone marrow / stem cell transplantation in children with recurrent malignant gliomas, medulloblastoma and ependymoma have been disappointing with significant morbidity and mortality. Intraoperative radiation has also been utilized for the treatment of primary and recurrent brain tumors. In a report from Japan, 17 patients including two children with radiation recurrent malignant brain tumors were treated with intraoperative radiation to doses of 20 - 40 Gy. Intraoperative radiation was delivered using special applicators and electron beams. The radiation was delivered after tumor resection and doses of 23 - 40 Gy were delivered to depths of 0.5-1.5 cm. The median survival for patients with malignant gliomas and other tumors (ependymoma, oligodendroglioma) was 12 months and 51 months respectively. The two children with ependymoma were cured and are currently alive at 134 and 88 months after intraoperative radiation. Three patients developed symptomatic brain necrosis, two of them had relief of symptoms with surgery and one patient died. Three patients also developed postoperative meningitis. In another report from University of Nebraska Medical Center, 49 patients with glioblastoma multiforme were treated with interstitial Cobalt 60 high dose-rate irradiation to a dose of 20 Gy to the tumor with a 1-cm margin. The patients with no prior radiation therapy (Group I) received an additional 40 Gy of external irradiation. Nineteen of these patients (Group II) had been previously irradiated, and they received only interstitial irradiation. The Cobalt 60 probe was guided into the tumor using CT scans and a stereotactic frame. This treatment was well tolerated, one patient had a dural leak and another had a subdural hematoma. There were no cases of meningitis or radiation necrosis. The median survival for Group I and Group II patients were 7 months and 6 months respectively.

The photon radiosurgery system (PRS) is an intraoperative irradiation device that is capable of delivering high radiation doses to brain tumors. This system has recently been approved for clinical use by the Food and Drug Administration (FDA).

Photon Radiosurgery System (PRS)

The Photon Radiosurgery System (PRS) incorporates a miniature, 40 KeV x-ray source capable of delivering a prescribed radiation dose directly to a target volume. The PRS consists in part of an electron beam-activated x-ray source with a sealed vacuum tube that is 10 cm long and 3.2 mm in outer diameter that is designed for insertion into the body. This vacuum tube incorporates an electron beam target on the inside surface of its tip. When an accelerated electron beam is generated and sent down the tube to strike the target, Bremsstrahlung and line x-rays are emitted from the tip of the tube in a nearly isotropic pattern.

Measurements of dose-rate in a water phantom have determined that the x-ray beam emanates essentially, from a point source, with a nominal dose rate of 150 cGy/min at 10 mm, for a beam current of 40 uA and a voltage of 40 kV. The absolute dose is estimated to be + 10%. The dose distribution in water falls off approximately as a function of the third power of the distance from the power source. The generator is light weighed, only 3.45 lbs. The radiation dose is adjusted by accelerating voltage (ranging from 30 to 50kV), beam current (ranging from 5 to 40 uA) and treatment time (0-60 minutes) through the control console that weighs only 40lbs. The lightweight of PRS system readily allows us to carry the device to the laboratory and the operating room.

For use of the PRS as an adjuvant treatment, treatment applicators made from a rigid biocompatible plastic (ULTEM 1000) with known x-ray transmission characteristics are used. The inside is hollowed out to allow introduction of the PRS x-ray probe to the epicenter of the applicator so that the dose at its outer surface is uniform. The end of the applicators is spherical with its diameter ranging from 1.5 cm to 4 cm. Treatment applicators will be sterilized prior to each use. The applicator is inserted into the tumor-resected cavity to deliver the prescribed dose of radiation.

The operation and dose characteristics of the PRS combine advantages of external beam radiosurgery with those of brachytherapy (implantation of radiation seeds). As with brachytherapy, the PRS can be located very precisely within the target volume, and can improve the delivery of conformal therapy by irradiating the target volume precisely, with little or no scatter of radiation. Due to its very rapid dose fall-off, the PRS significantly reduces the radiation dose delivered to healthy tissues as compared with external beam radiation and radiosurgery. Like radiosurgery, however, the PRS has a very high dose rate and can deliver high radiation doses to the target volume. Another distinct advantage of the PRS system is the ability to significantly decrease the radiation dose to the normal structures in the brain adjacent to the tumor. All of the radiation treatment techniques presently available deliver 10-50% of prescribed dose to the normal brain. Intraoperative irradiation using PRS because of its direct application into the tumor or tumor bed limits the dose to the normal tissue. This approach could result in a significant decrease in radiation induced complications in vital structures such as the optic pathway, brain stem and cerebral blood vessels. Another advantage of PRS is that unlike other types of therapy, the PRS does not require the use of a radiation-shielded room. To summarize, the advantages of the interstitial/surface application of radiation using the PRS are:

1. Direct access to the surgical bed of the tumor
2. Accurate delivery of a high single dose of radiation to the tumor
3. Superior protection of adjacent brain, cranial nerves or other critical structures by the use of intraoperative shielding or intraoperative displacement of these organs
4. Superior radiobiological effectiveness (RBE) of low energy X-rays
5. Tumor dose inhomogeneity similar to brachytherapy and Gamma knife radiosurgery, with the center of the tumor receiving a higher dose than the peripheral region that is adjacent to normal structures.

Results of studies carried out with the PRS in brain tumors have demonstrated it to be capable of delivering a lethal dose of radiation, in a single application to intracranial tumors with minimal side effects. It has been used to treat primary and metastatic brain tumors. In a report from Massachusetts General Hospital, 14 adults with primary and metastatic brain tumors < 3.5 cm in greatest diameter were treated with a single fraction of irradiation using PRS. The treated tumor diameter ranged from 10mm - 35 mm (mean 21mm), and the tumor edge prescribed dose ranged from 10-20 Gy (average 12.5 Gy). The average treatment time was 23 minutes (range, 7-45 minutes). Local control was obtained in 10 of the 13 patients with a follow-up of 1.5 - 36 months (mean 12 months). All patients tolerated the procedure well, and most patients were discharged home the day after treatment. No new neurological deficits were noted after irradiation. This study aims at determining the maximum tolerated dose of irradiation using PRS in recurrent pediatric brain tumors.

Dose Selection

The radiation dose delivered by the PRS and radiosurgery are similar with regard to dose-rate and total dose. The RTOG (Radiation Therapy Oncology Group) has performed a dose escalation study to assess the maximum tolerated dose of radiosurgery in adults with previously irradiated brain tumors and brain metastases. Based on acute and late toxicity, the maximum tolerated radiosurgery doses were 24 Gy, 18 Gy and 15 Gy for tumors < 20 mm, 21-30 mm and 31-40 mm respectively.

In this study we had intended to perform a similar dose escalation study with doses ranging from 10-19 Gy, 10-16 Gy and 10 - 14 Gy for tumors < 20 mm, 21-25 mm and 26-40 mm respectively. These doses are lower than the established maximum tolerated doses for brain reirradiation in adults with radiosurgery. These doses are also lower than the 20-40 Gy doses utilized for intraoperative irradiation of adult brain tumors with electrons and Cobalt 60 sources.

An interim analysis of patients entered on the study was performed. Based on the occurrence of treatment -related complications in ONE patient who required 2 applicators and in another patient in whom the dose was prescribed to 5 mm depth, the protocol has been modified as follows:

1. No patient will have PRS treatment using more than one applicator
2. The depth of prescribed dose should not exceed 2 mm
3. Patients who have received prior RT and those who have not received prior RT would be classified into Group A and Group B respectively.
4. The dose levels will for these two groups would be as shown in the table in Section 8.0. The dose escalation for non-brainstem (10-19 Gy) remains the same, but dose escalation will no longer be stratified by tumor size. The dose levels for sites adjacent to the brainstem and/or cranial nerves (10-14 Gy) also remain the same. A minimum of 3 patients will have to be accrued in each dose level and only if there are no complications observed, accrual at the next dose level would begin.

Dose escalation will be based on the incidence of acute CNS toxicity defined by RTOG criteria. Unacceptable toxicity will be considered to be irreversible grade 3 (severe), any grade 4 (life threatening) or grade 5 (fatal) RTOG CNS toxicity occurring within 3 months of reirradiation. If no patient developed an unacceptable CNS toxicity as defined below, the dose for that tumor size was then escalated.

The brain stem is very important part of the brain that controls most bodily functions like blood pressure, respiration etc. In this study, we have adopted a gentler dose escalation scheme for tumors in and around the brain stem. The three doses to be studied for tumors in this location are10 Gy, 12 Gy and 14 Gy. These doses will be delivered independent of tumor size.

ELIGIBILITY:
Inclusion Criteria:

* All patients must be between 2 and 32 yrs. of age. Patients who are pregnant or lactating will not be included in this study.
* Patients must have an estimated survival time of > 3 months, and a Karnofsky performance status of > 50% or and ECOG performance status of 0-2.
* Patient must have radiographic imaging evidence of tumor recurrence except for glioblastoma multiforme.
* The recurrent tumor prior to irradiation with PRS must be < 4 cm.
* All patients must be > 3 weeks from cytotoxic chemotherapy, except if patient received < 1 week of non-myelotoxic chemotherapy. In that case, patient may be enrolled with permission of the principal investigator.
* All patients must be > 6 weeks from high dose chemotherapy with stem cell rescue.
* All patients must be > 3 weeks from prior radiation therapy.
* Patients with a history of prior irradiation will be included.
* Informed consent must be obtained prior to registration on the study.

Tumor Sites:

* Brain
* Spinal Cord

Tumor Types:

* Recurrent Medulloblastoma
* Recurrent Ependymoma (recurrence regardless of primary treatment)
* Recurrent Glioma
* Glioblastoma Multiforme
* Recurrent Craniopharyngioma
* Recurrent PNET (Primitive Neuroectodermal tumor)
* Recurrent Meningioma
* Recurrent Pineoblastoma

Tumor Size:

* < 4 cm in maximum diameter

Ages: 2 Years to 32 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Estimated)
Dates: Start 2001-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose of radiation that can be delivered using the Photon Radiosurgery System (PRS) in children with radiation recurrent brain tumors. | End of study
To determine the maximum tolerated dose of radiation that can be delivered with a combination of external irradiation and radiosurgery using PRS in children with glioblastoma multiforme and children with recurrent ependymoma | End of study
To determine the tumor response following reirradiation with PRS. | End of study

SECONDARY OUTCOMES:
To determine the quality of life of children following irradiation with PRS. | End of study
To study gene expression in tumors before and after irradiation with PRS | End of study

CONTACTS AND LOCATIONS:
Overall Officials: Tadanori Tomita, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago; John A. Kalapurakal, MD, Principal Investigator — Northwestern Memorial Hospital
Locations (1):
- Children's Memorial Hospital, Chicago, Illinois, United States